CLINICAL TRIAL: NCT03682822
Title: Comparative Effectiveness of Routine Early Versus Delayed Amniotomy for Pregnancies Less Than 37 Weeks Gestational Age: A Randomized Open Label Trial (CEREAL)
Brief Title: Routine Early vs Delayed Amniotomy for Preterm Pregnancies: A Randomized Open Label Trial
Acronym: Cereal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Clifton O'Neill Brock, Clinical Fellow OBGYN, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0511
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Labor, Premature
Keywords: Pregnancy; labor induction; preterm
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early artificial rupture of membranes (Experimental): Women in this arm will undergo artificial rupture of membranes before 4 cm of cervical dilation is reached during induction of labor as long as the procedure is deemed clinically safe and feasible.
  Interventions: Procedure: Early Artificial rupture of membranes
- Delayed artificial rupture of membranes (Active Comparator): Women in this arm may undergo artificial rupture of membranes performed only after 4 cm of cervical dilation is reached during induction of labor. Rupture may also be performed after 10 hours of oxytocin administration with no cervical change.
  Interventions: Procedure: Delayed Artificial rupture of membranes

INTERVENTIONS:
Procedure: Early Artificial rupture of membranes — Women in this arm will undergo artificial rupture of membranes before 4 cm of cervical dilation is reached during induction of labor as long as the procedure is deemed clinically safe and feasible.
  Arms: Early artificial rupture of membranes
Procedure: Delayed Artificial rupture of membranes — Women in this arm may undergo artificial rupture of membranes performed only after 4 cm of cervical dilation is reached during induction of labor. Rupture may also be performed after 10 hours of oxytocin administration with no cervical change.
  Arms: Delayed artificial rupture of membranes

SUMMARY:
To compare the duration of preterm induction of labor in women undergoing early vs. late or no artificial rupture of membranes (AROM). Maternal and neonatal outcomes will also be compared between the two groups.

DETAILED DESCRIPTION:
Women presenting with a preterm singleton pregnancy between 28.0 and 36.6 weeks of gestation with cephalic lie and a medical indication for induction of labor will be approached for this study. The patient/provider must be attempting induction with the goal of vaginal delivery. Women with ruptured membranes, suspected intrauterine infection, prior uterine scar, fetal demise, or a fetal anomaly will be excluded. Women that agree to the study will be randomized to 2 groups: the "early amniotomy" group and the "late amniotomy" group.

Women in the early amniotomy group will undergo artificial rupture of membranes (AROM) prior to reaching cervical dilation of 4 cm. Women in the late amniotomy group may not undergo AROM until they reach cervical dilation of greater than 4 cm or they have been on an oxytocin drip for greater than 10 hours with no cervical change. It is possible that a woman in the late amniotomy group will not undergo AROM at all.

The primary outcome under consideration is time in labor. Secondary outcomes include rates of chorioamnionitis, postpartum endometritis, mode of delivery, and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Preterm singleton pregnancy between 28.0 and 36.6 completed weeks of gestation
* Fetus in the cephalic position
* Intent to induce labor for vaginal delivery
* If cervical ripening is planned, patient must be enrolled within an hour of initiation of ripening. If no ripening is planned, enrollment must be complete prior to starting induction.

Exclusion Criteria:

* Preterm premature rupture of membranes (PPROM)
* Fever or suspected chorioamnionitis prior to start of IOL
* Prior uterine scar
* Infection with HIV/Hepatitis B Virus (HBV)/Hepatitis C Virus (HCV) or an active Herpes Simplex Virus (HSV) infection
* Intrauterine fetal demise
* Major fetal anomaly
* Cervical dilation > 4 cm

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-22 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Total duration of labor. | Induction of labor until delivery (1 hr - 48 hrs)
  The duration of labor begins with administration of the first induction agent (i.e. Cook balloon, Foley catheter, prostaglandins, or oxytocin) and ends with delivery.

SECONDARY OUTCOMES:
Labor Outcomes:Time from completion of cervical ripening to delivery | Induction of labor until delivery (1 hr - 48 hrs)
  When the last induction agent is a foley/Cook balloon, or cervidil (dinoprostone), "completion of cervical ripening" will be defined as the time when the agent is removed. When the last induction agent is misoprostol, "completion of cervical ripening" will be defined as 4 hours after administration of the last dose.
Labor Outcomes: Delivery before 24 hours from start of Induction of Labor (IOL) | Induction of labor until delivery (1 hr - 48 hrs)
  A dichotomization of duration of labor
Labor Outcomes: Duration of the 2nd stage of labor | Induction of labor until delivery (1 hr - 48 hrs)
  Defined as time from the first cervical exam with complete dilation and effacement to the time of delivery
Maternal Outcome:Cesarean delivery | at delivery
  Mode of delivery
Maternal/Labor Outcomes: Indication for Cesarean delivery | at delivery
  Reason for cesarean delivery
Maternal/Labor Outcomes:Operative vaginal delivery | at delivery
  Use of either a vacuum device or obstetrical forceps
Maternal intrapartum fever or chorioamnionitis | during labor to delivery
  Defined as persistent intrapartum fever and/or suspected or confirmed intraamniotic infection (20)
Post-partum endometritis: | up to 10 days
  defined as postpartum febrile morbidity in the absence of another causative factor (i.e. wound infection, deep venous thrombosis). Postpartum febrile morbidity is defined as oral temperature ≥ 38.0⁰ C on any 2 of the first 10 days postpartum, exclusive of the first postpartum day
Epidural anesthesia | during labor
  Use of epidural regional anesthesia for pain control during induction of labor
Recurrent variable or late decelerations | during labor
  As defined by The American College of Obstetrics and Gynecology ( ACOG), practice bulletin No 110
Meconium stained amniotic fluid | during labor and delivery
  Meconium is noted in the amniotic fluid after rupture of membranes
Tachysystole | during labor
  As defined by ACOG, practice bulletin No 110
Use of amnioinfusion | during labor
  Placement of an intrauterine catheter and infusion of saline into the uterus during induction of labor
Use of intrapartum tocolytics | during labor
  Administration of a tocolytic drug during labor

CONTACTS AND LOCATIONS:
Overall Officials: Clifton O Brock, MD, Principal Investigator — University of Texas Health Science Center of Houston
Locations (1):
- University of Texas Health Science Center of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No